CLINICAL TRIAL: NCT01274611
Title: Comparing the Efficacy Between Suction-Curettage and Botox Injections in the Treatment of Axillary Hyperhidrosis
Brief Title: Botox and Suction-Curettage for Treatment of Excessive Underarm Sweating (Axillary Hyperhidrosis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU40780
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Axillary Hyperhidrosis
Keywords: sweating; sweat; underarm; axillary; hyperhidrosis; botox; liposuction; suction-curettage; suction; curettage
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A; Vacuum Curettage; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suction-Curettage (Active Comparator)
  Interventions: Device: Suction-Curettage
- Botox (Experimental)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botox will be injected into the underarm, targeting the sweat glands, to stop underarm sweating.
  Other Names: botox
  Arms: Botox
Device: Suction-Curettage — The doctor will insert a suction tool into two small incisions in order to suction out the sweat-producing glands. It is similar to liposuction, but instead of suctioning out fat, the doctor suctions out the layer of the deep skin where the sweat glands are located to decrease underarm sweating.
  Other Names: liposuction
  Arms: Suction-Curettage

SUMMARY:
The purpose of this study is to compare the effectiveness of two methods in the treatment of excessive underarm sweating (axillary hyperhidrosis): suction-curettage and Botox injections. Suction-curettage is a method in which the doctor will insert a suction tool into two small incisions in order to suction out the sweat-producing glands. It is similar to liposuction, but instead of suctioning out fat, the doctor suctions out the layer of the deep skin where the sweat glands are located. This method has been shown in some studies to effectively reduce underarm sweating for months at a time. Botox is a Food and Drug Administration (FDA) approved drug that in small doses, paralyses muscles. It is most commonly and famously used in the treatment of facial wrinkles. However, it has also been approved to treat excessive sweating. When injected in areas that sweat excessively, sweating can be significantly reduced in that area for months at a time. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65
* BMI 18.5 - 29.99
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies
* Subject is in good health
* Subject has the willingness and ability to understand and provide informed consent

Exclusion Criteria:

* Under age 18 or over age 65
* Pregnancy or lactating
* BMI ≥ 30 or ≤18.4
* Subjects who have undergone axillary suction/curettage any time in the past
* Subjects who have undergone axillary BT-A injections in the past year
* Subjects currently taking blood thinners or who have had chemotherapy or radiation within the last 6 months
* Subjects with a history of a bleeding disorder
* Subjects with an open, non-healing sore or infection near site of procedure
* Subjects with allergies to iodine, starch powder, albumin, or any botulinum toxin product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Onate, M.S., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from an urban, university based dermatology practice (Northwestern University, Chicago, IL) and the surrounding community. All patients provided written informed consent.
Pre-assignment Details: This was a split body, parallel-group randomized control trial with allocation ratio 1:1, using random block size of 2. The unit of randomization was the individual axilla.
Groups:
- Subjects Receiving Split Body Treatment: The unit of randomization was the individual axilla within each subject to receive either Botox treatment or suction-curettage treatment.
  Botox was injected into one underarm, targeting the sweat glands, to stop underarm sweating.
  For Suction-Curettage, the doctor inserted a suction tool into two small incisions in order to suction out the sweat-producing glands. It is similar to liposuction, but instead of suctioning out fat, the doctor suctions out the layer of the deep skin where the sweat glands are located to decrease underarm sweating.
Period: Overall Study
Arm/Group | Subjects Receiving Split Body Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was a parallel-group randomized control trial with allocation ratio 1:1, using random block size of 2. The unit of randomization was the individual axilla.
Groups:
- Subjects Receiving Split Body Treatment: The unit of randomization was the individual axilla within each subject to receive either Botox treatment or suction-curettage treatment.
  Botox wase injected into one underarm, targeting the sweat glands, to stop underarm sweating.
  For Suction-Curettage, the doctor inserted a suction tool into two small incisions in order to suction out the sweat-producing glands. It is similar to liposuction, but instead of suctioning out fat, the doctor suctions out the layer of the deep skin where the sweat glands are located to decrease underarm sweating.
Arm/Group | Subjects Receiving Split Body Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Secondary Outcome: The Change in Hyperhidrosis Disease Severity Scores From Baseline Compared to 3 Months After Treatment
Description: Change in mean score on the Hyperhidrosis Disease Severity Scale (HDSS) from baseline minus 3 months after treatment.
  The HDSS iquestionnaire assigns a point value to the patient's view:
  My sweating is...
  1. never noticeable and never interferes with my daily activities
  2. tolerable but sometimes interferes with my daily activities
  3. barely tolerable and frequently interferes with my daily activities
  4. intolerable and always interferes with my daily activities
  Lower point values are considered better and higher point values are considered worse.
  A larger change in score between baseline and 3 months is considered a better outcome and a smaller change in score is considered a worse outcome for each treatment. Change scores were calculated (baseline minus 3 months). Positive change scores indicate that scores were better; negative change scores indicate their scores were worse after treatment.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: axillae
Groups:
- Botox: Botox was injected into the underarm, targeting the sweat glands, to stop underarm sweating.
- Suction-Curettage: The doctor inserted a suction tool into two small incisions in order to suction out the sweat-producing glands. It is similar to liposuction, but instead of suctioning out fat, the doctor suctions out the layer of the deep skin where the sweat glands are located to decrease underarm sweating.
Arm/Group | Botox | Suction-Curettage
Number analyzed (Participants) | 20 | 20
Number analyzed (axillae) | 20 | 20
Scores on a scale | 1.55 (0.68633) | 0.08 (0.83351)
Statistical Analysis 1: Comparison: Botox vs Suction-Curettage; Test type: Non-Inferiority or Equivalence — A sample of 20 patients, or 40 treatment sites (the unit of randomization), provided 80% power to detect effect sizes of 0.68 using a paired t test at a type I error rate of 5%; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 0.80

2. Primary Outcome: Percentage Change of Sweat Rate (mg/Min) at Baseline Compared to 3 Months
Description: The primary outcome measure was the treatment associated unilateral axillary percentage change of sweat rate in milligrams per minute in the exercise-induced state measured at baseline compared with the sweat rate measured 3 months after treatment.
  This process entails placing filter paper on the area of concern for a specific amount of time, after which the paper is weighed and sweat production is quantified in units of weight per time. The amount of sweat produced was recorded in milligrams per minute by subtracting the initial weight of the paper segment before exercise from the final, post-application weight, after exercise and dividing by 5 minutes.
  Percentage sweat rate was calculated as [(sweat rate at baseline - sweat rate at 3 months)/sweat rate at baseline]*100 with a positive percent change indicating sweat rate reduction if the baseline had a higher sweat rate.
Time Frame: baseline and 3 months
Measure: Mean (Full Range); unit: Percentage Change
Units Other Than Participants: axillae
Arm/Group | Botox | Suction-Curettage
Number analyzed (Participants) | 20 | 20
Number analyzed (axillae) | 20 | 20
Percentage Change | 73.8 [20 to 100] | 58.8 [2 to 94]
Statistical Analysis 1: Comparison: Botox vs Suction-Curettage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.01, t-test, 2 sided; Mean Difference (Net) = 15

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Botox | Suction-Curettage
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
There was a the lack of long-term assessment of comparative effectiveness. It is uncertain whether suction-curettage removes the eccrine sweat glands or mainly the apocrine glands.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes